CLINICAL TRIAL: NCT01477515
Title: Endocannabinoids in End Stage Renal Disease
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Allon Friedman, Assistant Professor of Medicine, Indiana University
Other Study IDs: ANF-1
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: End Stage Renal Disease; Nutrition
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- End stage renal disease patient
- Matched controls

SUMMARY:
To investigate the relationship between dietary intake, body habitus, and endocannabinoid levels in end stage renal disease patients as compared to matched controls.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patient, able to give informed consent

Exclusion Criteria:

* hospitalization in past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients healthy control subjects
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-02